CLINICAL TRIAL: NCT00776126
Title: Radiologists' Preference Study - Digital Breast Tomosynthesis
Brief Title: Digital Breast Tomosynthesis Preference Study
Acronym: NRR
Status: Completed | Type: Observational
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: LCCC 0803
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2017-03-06 (Actual); Status verified 2017-03

CONDITIONS: Breast Cancer
Keywords: Breast; 3D Digital Mammography; Digital Breast Tomosynthesis
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: All enrolled subjects will undergo digital breast tomosynthesis.
  Interventions: Device: Digital Breast Tomosynthesis Exam

INTERVENTIONS:
Device: Digital Breast Tomosynthesis Exam — Digital Breast Tomosynthesis Exam consisting of single view (MLO) of each breast will be performed.

SUMMARY:
Mammography remains the current standard in the detection of breast cancer. However, conventional two-view mammography will not detect all cancers. The major limiting factor of conventional mammography is the presence of superimposed breast tissue that can obscure clinically significant lesions. It is this limitation that decreases the sensitivity of mammography and leads to false negative results.

The recent development of digital detectors has allowed imaging technologies such as tomosynthesis to become clinically feasible. The examination, similar to conventional mammography with regard to patient positioning and glandular dose, allows acquisition of a digital data set that can be reconstructed and viewed in multiple sections. The ability of tomosynthesis to unmask overlapping structures has been shown in preliminary studies to increase lesion visibility. Used as either a primary imaging modality, or as an adjunct to screening mammography, tomosynthesis has the potential to provide increased sensitivity and a lower number of false negative examinations.

The purpose of this study is to compare radiologist impression of digital breast tomosynthesis to digital mammography with respect to their ability to see and characterize specific lesion features.

ELIGIBILITY:
Inclusion Criteria:

* The subject is a woman ≥18 years of age or older who has no history of symptoms and/or physical signs of breast cancer in either breast (or, if she has had a mastectomy, in the remaining breast);
* The asymptomatic subject previously (within 3 months) underwent routine screening DM, which showed one or more abnormalities, and was referred for diagnostic mammography within the 30 days before study entry. The images from the screening examination must be available. If the prior screening examination was not conducted at the recruiting site, review of those images by the investigator must confirm that the recommendation for diagnostic mammography is warranted;
* The subject is able and willing to comply with study procedures, and has signed and dated the informed consent form;
* The subject is either surgically sterile (has had a documented bilateral oophorectomy and/or documented hysterectomy), or postmenopausal (cessation of menses for more than one year); or, if of childbearing potential, the possibility of pregnancy is remote based on a negative patient history or a negative urine pregnancy test.

Exclusion Criteria:

* The subject is pregnant or trying to become pregnant;
* The subject has been previously included in this study;
* The subject has a history of any symptoms and/or physical signs of breast cancer in either breast (or if she has had a mastectomy, no signs or symptoms of breast cancer in the remaining breast);
* The subject has breasts too large to be adequately positioned on 19 x 23 centimeter (cm) FFDM digital receptor without anatomical cut off during a DBT examination;
* The subject has participated in any of the on-going GE studies (GE 190-001, GE 190-002 or GE 190-003), or is participating in, or has participated in (within the prior 30 days), another trial of an investigational product;
* Has breast implant(s).
* Has reconstructed breast(s).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult women who have undergone previous screening with CR digital mammography and were scheduled for diagnostic workup with full-field digital mammography (FFDM).
Sampling Method: Non-Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2008-10; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Reader Preference | upon recruitment/enrollment phase completion

CONTACTS AND LOCATIONS:
Overall Officials: Amy S Campbell, MD, Principal Investigator — University of South Carolina; Etta D Pisano, MD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- Breast Imaging Clinic; University of North Carolina Hospitals, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Diekmann F, Bick U. Tomosynthesis and contrast-enhanced digital mammography: recent advances in digital mammography. Eur Radiol. 2007 Dec;17(12):3086-92. doi: 10.1007/s00330-007-0715-x. Epub 2007 Jul 28. PMID 17661053
- [Background] Gong X, Glick SJ, Liu B, Vedula AA, Thacker S. A computer simulation study comparing lesion detection accuracy with digital mammography, breast tomosynthesis, and cone-beam CT breast imaging. Med Phys. 2006 Apr;33(4):1041-52. doi: 10.1118/1.2174127. PMID 16696481
- [Background] Niklason LT, Christian BT, Niklason LE, Kopans DB, Castleberry DE, Opsahl-Ong BH, Landberg CE, Slanetz PJ, Giardino AA, Moore R, Albagli D, DeJule MC, Fitzgerald PF, Fobare DF, Giambattista BW, Kwasnick RF, Liu J, Lubowski SJ, Possin GE, Richotte JF, Wei CY, Wirth RF. Digital tomosynthesis in breast imaging. Radiology. 1997 Nov;205(2):399-406. doi: 10.1148/radiology.205.2.9356620.
- [Background] Poplack SP, Tosteson TD, Kogel CA, Nagy HM. Digital breast tomosynthesis: initial experience in 98 women with abnormal digital screening mammography. AJR Am J Roentgenol. 2007 Sep;189(3):616-23. doi: 10.2214/AJR.07.2231. PMID 17715109